CLINICAL TRIAL: NCT01237483
Title: A Phase II Study, Multicenter, to Evaluate the Efficacy and Safety of the Combination of Reirradiation - Erbitux in Subjects Previously Irradiated and With a Local Recurrent Inoperable Squamous Cell Cancer of the Head and Neck
Brief Title: Reirradiation and Erbitux in the HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2008-01
Record Dates: First submitted 2010-11-08; First posted 2010-11-09 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Head and Neck Cancer Squamous Cell
Keywords: reirradiation with Erbitux; HNSCC; local recurrent inoperable Squamous Cell Cancer of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erbitux Radiotherapy (Other): Radiotherapy during 5 weeks and concurrent Erbitux once a week.
  Interventions: Drug: Erbitux

INTERVENTIONS:
Drug: Erbitux — To begin 7 days before radiotherapy, loading dose 400 mg / m² in the first week then 250 mg / m² weekly for the duration of radiotherapy (for a total of 7 doses including the loading dose)

SUMMARY:
The purpose of this study is to investigate in patients with cancer of the throat and recurrent inoperable a different modality treatment consisting of radiation continuously for 5 weeks and half associated with a drug directed against a receptor on cell surfaces cancer, called Erbitux ®.

The investigators hope with this shorter treatment (1.5 weeks less than the usual treatment) to improve the antitumor efficacy without additional toxic side effects.

DETAILED DESCRIPTION:
We hope with this treatment improved antitumor efficacy without additional toxic side effects, while being shorter than 1.5 weeks of standard therapy. But this is an hypothesis we can not meet the current state of knowledge, which justifies this study.

The main hypothesis is that this combination of reirradiation and Cetuximab give a relative gain of 15% complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unresectable locoregional recurrence of squamous cell carcinoma in a previously irradiated area (at least 75% of the volume of recidivism must be in an area who have received at least 50 Gy)
* The entire tumor volume can be included in a radiation field without the total dose to the spinal cord more than 50 Gy (dose + dose earlier predicted)
* Patient with recurrent or second location in the oral cavity, oropharynx, larynx, hypopharynx, cervical lymph nodes or tissues, without distant metastases,
* Minimum 12 months after the end of radiotherapy previous
* WHO performance status: 0-1,
* Evaluable disease by RECIST V.1.1.,
* Age between 18 and 75 years
* The patient may have received prior chemotherapy for relapse for more than five weeks,
* The patient may have received cetuximab for the treatment of disease but not for the first relapse,
* Hematologic function: ANC ≥ 1500/mm3, Platelets ≥ 100000/mm3,
* Normal renal function: serum creatinine ≤ 120 µmol/l and/or creatinine clearance > 60 ml/min
* Normal liver function: bilirubin <1.5 x ULN, alkaline phosphatase and transaminases <2.5 x ULN,
* Normal cardiac function, assessed clinically. History of cardiovascular disease stabilized for over 12 months
* Cons-Lack of medical indications in the proposed treatment,
* The dosimetry of previous treatment should be available and the estimated dosimetry must be performed to check the constraints,
* All patients of childbearing age should receive effective contraception,
* Membership of a social security system (or be a beneficiary of such a plan) under the terms of the Act of August 9, 2004,
* Signed informed consent

Exclusion Criteria:

* Tumors of the nasal cavity and paranasal,
* Tumors of other histological type,
* Stage IV with distant metastases or multiple tumors,
* Time after previous radiotherapy <12 months,
* Less than 75% of the volume of relapse who have previously received at least 50 Gy,
* Any medical condition or general-cons would indicate the completion of treatment. Systemic disease or uncontrolled infection,
* History of cancer other than head and neck cancer, cutaneous basal cell, carcinoma in situ of the cervix
* Any other concurrent anticancer therapy,
* Patient receiving another molecule experimental
* Pregnant, lactating or without contraception;
* Persons deprived of liberty under guardianship
* Inability to undergo medical test for geographical, social or psychological
* Nasopharyngeal Neoplasms
* Patients with active ischemic heart disease or previous myocardial infarction within the last 12 months
* Late toxicity dermal or subcutaneous related to previous irradiation of grade> 2 in the scale CTCAE V.4.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
The main objective is to evaluate the complete response rate of the association re-irradiation - Erbitux ®. | It will be measured by spiral CT scan or magnetic resonance imaging (MRI), 2 months after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laurent MARTIN, oncologist, Study Director — Centre Guillaume Le Conquérant, 76600 Le Havre, France; Claude TUCHAIS, oncologist, Principal Investigator — Centre Paul Papin, 49933 Angers, France; Sauveur Marc ALFONSI, oncologist, Principal Investigator — Institut Sainte Catherine, 84082 Avignon, France; Xu Sh SUN, oncologist, Principal Investigator — Hôpital Jean Minoz, 25030 Besançon, France; Dominique DE RAUCOURT, oncologist, Principal Investigator — Centre François Baclesse, 14076 Caen, France; Michel LAPEYRE, oncologist, Principal Investigator — Centre Jean Perrin, 63011 Clermond-Ferrand, France; Philippe MAINGON, oncologist, Principal Investigator — Centre G-F Leclerc, 21079 Dijon, France; Muriel GARCIA-RAMIREZ, oncologist, Principal Investigator — Hôpital Robert Boulin, 33505 Libourne, France; Christian SIRE, oncologist, Principal Investigator — Hôpital du Scorff, 56322 Lorient, France; Séverine RACADOT, oncologist, Principal Investigator — Centre Léon Bérard, 69373 Lyon, France; Véronique FAVREL, oncologist, Principal Investigator — Centre Hospitalier Lyon Sud, 69495 Pierre-Benite, France; Etienne BARDET, oncologist, Principal Investigator — Centre René Gauducheau, 44805 Nantes-St Herblain, France; Philippe LANG, oncologist, Principal Investigator — Hôpital de La Pitié Salpitrière, 75013 Paris, France; Isabelle TENNEVET, oncologist, Principal Investigator — Centre Henri Becquerel, 76038 Rouen, France; Patricia BURBAN, oncologist, Principal Investigator — Clinique Armoricaine de Radiologie, 22015 St Brieuc, France; Olivier GALLOCHER, oncologist, Principal Investigator — Clinique Pasteur, 31300 Toulouse, France; Olivier GALLOCHER, oncologist, Principal Investigator — Polyclinique du Parc, 31078 Toulouse, France; Yungan TAO, oncologist, Principal Investigator — Institut Gustave Roussy, 94805 Villejuif, France; Pierre BOISSELIER, oncologist, Principal Investigator — Val d'Aurelle 34298 Montpellier cedex; Frédéric PEYRADE, oncologist, Principal Investigator — Centre Antoine Lacassagne 06189 NICE cedex 2; Marie SALIOU, oncologist, Principal Investigator — Clinique de l' Estuaire 44600 Pornichet; Cédrik LAFOND, oncologist, Principal Investigator — Centre Jean Bernard 72000 Le Mans; René-Jean BENSADOUN, oncologist, Principal Investigator — CHU 86021 Poitiers cedex; Alexandre COUTTE, oncologist, Principal Investigator — CHU Amiens sud 80004 Amiens; Hao QIU, oncologist, Principal Investigator — CHU 86000 Limoges; Florence HUGUET, oncologist, Principal Investigator — Hôpital Tenon 75020 Paris; Sébastien GUIHARD, Principal Investigator — Centre Paul Strauss 67065 Strasbourg; Xu Shan SUN, oncologist, Principal Investigator — Centre Hospitalier de Belfort Montbéliard Bd du Maréchal Juin 25200 Montbéliard
Locations (1):
- Hôpital Bretonneau, Tours, France